CLINICAL TRIAL: NCT00206492
Title: A Neoadjuvant Phase II Trial of ZD1839 (Iressa) and Tamoxifen in Inoperable Locally Advanced HER2-Overexpressing, ER-Positive Breast Cancer Patients: Biologic Correlative Study (AZ #1839US/0303)
Brief Title: Trial of ZD1839 (Iressa) and Tamoxifen in Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: halted by the PI only 3 of 45 subjects were accrued.
Sponsor: Baylor Breast Care Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H 13546
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Breast; Cancer; Neoadjuvant; HER2; Overexpressing
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Gefitinib; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iressa and Tamoxifen (Experimental): Iressa and Tamoxifen
  Interventions: Drug: Iressa; Drug: Tamoxifen

INTERVENTIONS:
Drug: Iressa — Iressa
  Other Names: ZD1839
Drug: Tamoxifen — Tamoxifen

SUMMARY:
The researchers want to learn whether ZD1839 can improve the activity of tamoxifen, a drug that participants will receive for the treatment of the type of breast cancer being studied. Tamoxifen medicine is part of the standard treatment for the type of breast cancer being studied. It is approved for the treatment of this problem. In order to help the researchers understand how the cancer responds to these medicines, the researchers will take a small tissue sample (biopsy) of the breast cancer before beginning treatment and after two weeks of treatment, at 6 weeks and when surgery is done as part of treatment for the cancer. If participants do not respond to treatment, another biopsy will be done to see why the participants did not respond. These samples will also be collected to look at different characteristics of the cancer. The researchers cannot and do not guarantee that participants will benefit if they take part in this study

DETAILED DESCRIPTION:
Epidermal growth factor receptor (EGFR) is expressed or over-expressed in many human solid tumors and plays an important role in progression to invasion and metastases. The EGFR tyrosine kinase is activated by binding of a variety of ligands to the external domain. Autophosphorylation by the EGFR tyrosine kinase initiates a signaling cascade that feeds downstream cell cycle control machinery regulating cell proliferation, and these reactions are a major component in growth factor-induced proliferation of cancer cells.

The Erb-B (HER) receptor family consists of four transmembrane tyrosine kinases: Erb-B1-epithermal growth factor receptor (EGFR, HER1), Erb-B2/neu (HER2), Erb-B3 (HER3), and Erb-B4 (HER4). The ectodomain of Erb-B1, Erb-B3, and Erb-B4 interacts with a specific set of ligand, whereas no ligand has been identified thus far for the Erb-B2 receptor. Nonetheless, Erb-B2 can be activated by any of the other ligand-activated Erb-B coreceptors. Upon ligand binding to the active domain of Erb-B1, Erb-B3, or Erb-B4, these receptors preferentially recruit Erb-B2 into a heterodimeric complex in which the Erb-B2 kinase can modulate receptor internalization and prolong signal transduction.

Data are now emerging that Erb-B2 modulates cellular p27 and cyclin D1 protein levels through both Ras/MAP kinase and PI3K/Akt signaling. Reversible interruption of Erb-B2 function by trastuzumab (Herceptin) has been shown to inhibit MAPk and reduce MAPk-mediated transcription through cyclin D1. In addition, the signaling molecule Akt is important in the cell survival pathway. Akt inhibits apoptosis and is present in the PI3 kinase pathway, which is activated by the EGF family and the IGF family. Several biologic arguments support the use of EGR inhibitors to block HER2 signaling. In HER2-overexpressing cell lines, the HER2 receptor is constitutively phosphorylated. This suggests that HER2 may be transactivated through ligand-stimulated EGFR, also present in tumor cells. In addition, overexpression of HER2 enhances the binding of EGFR ligands to the receptor and potentiates EGFR signaling. HER2 inactivation has been shown to impair EGFR- mediated transformation, and conversely EGFR blocking antibodies can augment the growth inhibitory effect of antiHER2 antibodies in cells with high levels of HER2. Taken together, these data suggest that EGFR/HER2 crosstalk is present in a subset of human tumors and that interruption of EGFR may reduce HER2 signaling. Cell cycle progression is regulated predominantly by cyclin-dependent kinases (CDKs), which in turn are controlled by a family of CDK inhibitory proteins that include P27KIP1 and P21CIP1-WAF1. Pathways involving CDK inhibitors are commonly destructive in cancer cells. ZD1839 is an orally active, selective EGFR tyrosine kinase inhibitor that blocks signal transduction pathways implicated in cancer cell proliferation, survival, and other host-dependent processes promoting cancer growth.

In preclinical studies, ZD1839 causes tumor growth delay in a range of cancer cell lines and xenografts, and tumor regression has been observed at higher doses. ZD1839 was also shown to inhibit proliferation in DCIS together with significantly increased apoptosis in these tissues. Data from these different cell lines and xenografts suggest that ZD1839 may act via dose-dependent growth inhibition and by increasing apoptosis, and may even potentiate the activity of cytotoxic chemotherapy.

In one phase II multicenter study, 63 women with metastatic breast cancer who could have had any number of previous chemotherapy or hormonal regimens were treated with an oral daily dose of 500 mg of ZD1839 until disease progression, intolerable toxicity, or withdrawal of consent. Dosage reduction to 250 mg daily was allowed for toxicity. The primary end point was clinical benefit rate (complete response + partial response [modified ICC/WHO criteria] + stable disease) at 6 months. There was 1 partial response and 2 patients with stable disease for more than 4 months (4 months in 1 patient and 7+ months in the other), for a total of 4.8% clinical benefit. An additional 4 patients had stable disease lasting 1 to 2 months, and another 2 patients had stable disease lasting 1 month, resulting in an overall 14.3% partial response or stable disease in this heavily pre-treated population; 15% were on treatment for 4 to 8+ months, and 2 patients stayed on treatment, despite progression, because of significant bone pain palliation.

Preliminary efficacy and toxicity data from another phase II trial of 22 ER-positive or ER-negative patients were reported at the same conference. In that study, patients could have had 1 previous chemotherapy regimen or were experiencing disease progression while on tamoxifen and were given 500 mg of ZD1839 daily. Two patients had a partial response and 10 had stable disease at 4 weeks. In both trials the toxicity profile was identical to that seen in patient with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be female and must have signed an informed consent form.
2. Primary breast cancers must be human epidermal growth factor receptor (HER2) overexpressing (2+ or 3+, or both, as determined by immunohistochemistry [IHC]), and estrogen receptor (ER) positive. Primary breast cancers must be of clinical and/or radiologic size >4 cm, with or without gross metastatic disease according to the International Union against Cancer (UICC) modified World Health Organization (WHO) criteria.
3. Negative serum pregnancy test (bHCG) within 7 days of starting study, if of child-bearing potential.
4. Adequate bone marrow function:

   * Hematocrit >30%,
   * total neutrophil count must be >1.5 x 10^9/L, and
   * platelet count >100 x 10^9/L.
5. Renal function tests:

   * creatinine within 1.5 times the institution's upper limit of normal (ULN).
6. Liver function tests:

   * Total serum bilirubin within ULN,
   * liver transaminases within 2.5 x ULN,
   * alkaline phosphatase within 5 x ULN.
7. Performance status (WHO scale) <2.
8. Age > 18 years.

Exclusion Criteria:

1. Pregnancy or unwillingness to use a reliable contraceptive method in women of child-bearing potential.
2. Women who are lactating or breastfeeding.
3. Severe underlying chronic illness or disease.
4. Patients on other investigational drugs while on study will be excluded.
5. Severe or uncontrolled hypertension, history of congestive heart failure, acute myocardial infarction, or severe coronary arterial disease.
6. No previous or current malignancies at other sites within the preceding 5 years, with the exception of adequately treated, cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
7. Any evidence of ongoing interstitial lung disease.
8. Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort.
9. Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
10. Known severe hypersensitivity to ZD1839 or any of the excipients of this product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-07; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
cellular response | 10 years
  mechanisms of the cellular response, markers predicting response, by investigating whether ZD1839 with or without tamoxifen treatment is associated with altered biomarkers in cells isolated by core needle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — Baylor Breast Center
Locations (1):
- Baylor Breast Center, Houston, Texas, United States

REFERENCES:
- See also: Web site — http://www.breastcenter.tmc.edu